CLINICAL TRIAL: NCT05797506
Title: Safety, Feasibility and Efficacy of Sulforaphane (Avmacol Extra Strength) in Chronic Kidney Disease - Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Safety, Feasibility and Efficacy of Sulforaphane (Avmacol Extra Strength) in Chronic Kidney Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: University of Virginia (Other); Nutramax Laboratories, Inc. (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Thu Le, John J. Kuiper Distinguished Professor of Medicine & Chief, Division of Nephrology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00008014; R01DK128677 (NIH)
Record Dates: First submitted 2023-03-02; First posted 2023-04-04 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Disease Stage 3; Chronic Kidney Disease Stage 4
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — sulforaphane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sulforaphane (Avmacol Extra Strength) (Experimental): Four tablets of Sulforaphane (Avmacol Extra Strength) per day. The tablets will be provided by Nutramax.
  Interventions: Drug: Sulforaphane (Avmacol Extra Strength)
- Placebo (Placebo Comparator): Nutramax will provide the matched placebo tablets.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Sulforaphane (Avmacol Extra Strength) — 4 Tablets of Sulforaphane (Avmacol Extra Strength) per day in patients with Chronic Kidney Disease, stages 3-4.
  Arms: Sulforaphane (Avmacol Extra Strength)
Dietary Supplement: Placebo — These tablets will be matched placebos and will be provided by Avmacol.
  Arms: Placebo

SUMMARY:
The Sulforaphane Production System® in Avmacol Extra Strength (ES) supplies broccoli seed extract (glucoraphanin) and Myrosimax® (Active Myrosinase Enzyme) which helps promote sulforaphane production in your body. The investigators hypothesize that daily intake of Avmacol ES can decrease kidney disease progression rate and decrease markers of oxidative stress and inflammation in Chronic Kidney Disease (CKD) patients. They will test this hypothesis in a randomized, double-blind, placebo controlled Phase 2 clinical trial. This proposed study has been funded by the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), R01 DK128677.

DETAILED DESCRIPTION:
The investigators will test the safety and efficacy of Avmacol ES in Chronic Kidney Disease (CKD) patients. After having established a safe dose of 4 tablets once daily in participants with CKD Stages 3 - 4 in the pharmacokinetic (PK) phase, the investigators will enroll 100 participants from the Kidney Clinic at the University of Rochester Medical Center and Highland Hospital with CKD stages 3 - 4 who will be randomized to Avmacol ES or placebo in a 1:1 ratio in a blinded manner.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 80 years
* Estimated glomerular filtration rate (eGFR) ≥ 20 and < 60 mL/min/1.73m2 and a decline in eGFR of ≥ 3 ml/min/1.73m2 /year in the previous 12 ± 2 months
* Able to provide consent
* Able to swallow Avmacol ES or placebo capsules

Exclusion Criteria:

* Significant co-morbid conditions with life expectancy of < 1 year
* Serum potassium of > 5.5 milliequivalents per liter (mEq/L) at screening
* New York Heart Association Class 3 or 4 heart failure symptoms, known Ejection Fraction (EF) ≤ 30% or hospital admission for heart failure within the past 3 months
* Factors judged to limit adherence to interventions based on appointment attendance and medication treatment compliance; PI will make this determination
* Current participation in another medical intervention study
* Known to be pregnant or planning to become pregnant or currently breastfeeding; determined by self-report and medical record history. A urine pregnancy test will be completed for individuals of childbearing potential before administering the study drug, and repeated thereafter at every study visit (~ every 3-4 months)
* History of dementia documented in the medical record
* On anticoagulants or immunosuppression
* Under treatment for cancer
* Delayed gastric emptying or similar GI conditions Non-English-speaking individuals are excluded in this randomized phase of the study because the lack of English proficiency will affect a subject's ability to report problems or adverse events. If a patient cannot read, the consent form will be read to them by the research coordinator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal change in the scores | Seven timepoints per patient (baseline; month 1; month 2; month 3; month 4; month 5, and month 6)
  Patient-Reported Outcomes Measurement Information System (PROMIS®) Scale v1.2 - Global Health questionnaire. Scoring: The questionnaire has two scores: Physical Health (physical health, physical function, pain, and fatigue items) and Mental Health (quality of life, mental health, satisfaction with discretionary social activities, and emotional problem items). In all cases, a high score means more of domain. T scores for both Physical and Mental Health scales. In all cases, a high score means more of domain. For example, higher scores on physical functioning measure indicate better health.
Longitudinal change in the scores | Seven timepoints per patient (baseline; month 1; month 2; month 3; month 4; month 5, and month 6)
  Modified Kansas City Cardiomyopathy questionnaire (KCCQ) - All KCCQ scores are scaled from 0 to 100. A higher score indicates better health status.
Longitudinal change in the scores | Seven timepoints per patient (baseline; month 1; month 2; month 3; month 4; month 5, and month 6)
  Patient-Reported Outcomes Measurement Information System (PROMIS®) Scale v1.0 - Gastrointestinal Belly Pain 5a questionnaire. The PROMIS GI measures use a T-score centered on the U.S. General Population. This means that a score of 50 represents the average of the general population (and that 10 represents the standard deviation). A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like belly pain, a T-score of 60 is one SD worse than average. By comparison, a gastrointestinal symptom T-score of 40 is one SD better than average.
Longitudinal change in both systolic and diastolic blood pressure | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - millimeters of mercury (mmHg)
Longitudinal change in 8-isoprostane in plasma | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - picograms per milliliter (pg/mL)
Longitudinal change in 8-isoprostane in urine | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - picograms per milliliter (pg/mL)
Longitudinal change in urinary albumin | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - μg/ml
Longitudinal change in protein/creatinine ratio | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - milligram per gram (mg/g)
Longitudinal change in plasma hydrogen sulfide | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - Nanomolar (nM)
Longitudinal change in plasma interleukin-6 | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - picograms per milliliter (pg/mL)
Longitudinal change in urine nephrin | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - microgram per milliliter μg/mL
Longitudinal change in messenger RNA (mRNA) levels of cytoprotective enzymes in peripheral blood mononuclear cells (PBMCs) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - Relative copy number
Longitudinal change in messenger RNA (mRNA) levels of heat shock proteins in peripheral blood mononuclear cells (PBMCs) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - Relative copy number
Longitudinal change in sodium as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - Millimoles per liter (mmol/L)
Longitudinal change in potassium as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - Millimoles per liter (mmol/L)
Longitudinal change in chloride as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - Millimoles per liter (mmol/L)
Longitudinal change in carbon Dioxide as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - Millimoles per liter (mmol/L)
Longitudinal change in anion Gap as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - milliequivalents per liter (mEq/L)
Longitudinal change in blood urea nitrogen as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - Milligrams per decilitre (mg/dL)
Longitudinal change in creatinine as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - Milligrams per decilitre (mg/dL)
Longitudinal change in estimated Glomerular Filtration Rate (eGFR) as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - milliliters of cleansed blood per minute per body surface (mL/min/1.73m2)
Longitudinal change in calcium as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - Milligrams per decilitre (mg/dL)
Longitudinal change in total protein as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - Grams Per Deciliter (g/dL)
Longitudinal change in albumin as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - Grams Per Deciliter (g/dL)
Longitudinal change in total bilirubin as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - Milligrams per decilitre (mg/dL)
Longitudinal change in aspartate transaminase (AST) as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - units per liter (U/L)
Longitudinal change in alanine transaminase (ALT) as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - units per liter (U/L)
Longitudinal change in alkaline phosphatase (ALP) as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - units per liter (U/L)
Longitudinal change in phosphorus as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - Milligrams per decilitre (mg/dL)
Longitudinal change in glucose as part of comprehensive metabolic panel (CMP) | Four timepoints per patient (baseline, month 1, month 3, and month 6)
  Unit of measurement - Milligrams per decilitre (mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No